CLINICAL TRIAL: NCT03959748
Title: DataBase of pulmoNary hyPertesion in PoLish Population - BNP-PL
Acronym: BNP-PL
Status: Recruiting | Type: Observational
Sponsor: Polish Cardiology Association (Other)
Collaborators: Jagiellonian University (Other)
Responsible Party: Sponsor
Other Study IDs: 1/BNP-PL/2018
Record Dates: First submitted 2019-03-26; First posted 2019-05-22 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension; Pulmonary Arterial Hypertension
Keywords: Pulmonary Hypertension,; CTEPH; Pulmonary Arterial Hypertension; Registry; Data Base; Polish patients
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PAH adults: Patients with pulmonary arterial hypertension who are at least 18 years old at study entry
- PAH children: Patients with pulmonary arterial hypertension who are at least 3 months old and are less than 18 years old at study entry
- CTEPH: Patients with chronic thromboembolic pulmonary hypertension who are at least 18 years old at study entry

SUMMARY:
The BNP-PL is a multicenter, observational study in which patients are prospectively followed in order to investigate clinical course and management of pulmonary hypertension in Poland.

All patients diagnosed with pulmonary arterial hypertension and chronic thromboembolic pulmonary hypertension confirmed in right heart catheterization, will be eligible to participate in the study.

DETAILED DESCRIPTION:
The BNP-PL Registry is an initiative of the Polish Cardiac Society Task Force for Pulmonary Vascular Diseases This study is conducted by the Polish Cardiac Society. All centers of pulmonary hypertension in Poland which are accredited by the National Health Fund have been invited to join the study. The data is administrated by the Jagiellonian University Medical College on the basis of an agreement between the Polish Cardiac Society, Jagiellonian University Medical College and pulmonary hypertension centres.

The goal is to describe current practice and outcomes in patients with pulmonary arterial hypertension and chronic thromboembolic pulmonary hypertension.

The data collection will have no impact on the way the patient is diagnosed and treated.

Collection of data on patients with pulmonary hypertension is carried out via the electronic platform.

No personal data is entered into the project database.

ELIGIBILITY:
Inclusion Criteria:

Patients with pulmonary arterial hypertension or chronic thromboembolic pulmonary hypertension diagnosed after 1st March 2018 (incident cases) who:

* are aged > 3 months at the time of enrollment
* fulfill the following hemodinamic criteria: mean pulmonary arterial pressure (mPAP) of 25 mm Hg or more, mean pulmonary arterial wedge pressure (PAWP) or left ventricular end-diastolic pressure (PVEDP) of 15 mm Hg or less, pulmonary vascular resistance (PVR) of 3 Woods.

Patients with pulmonary arterial hypertension or chronic thromboembolic pulmonary hypertension diagnosed before 1st March 2018 (prevalent cases) who:

* are aged > 3 months at the time of enrollment
* fulfill the following hemodinamic criteria: mean pulmonary arterial pressure (mPAP) of 25 mm Hg or more, mean pulmonary arterial wedge pressure (PAWP) or left ventricular end-diastolic pressure (PVEDP) of 15 mm Hg or less, pulmonary vascular resistance (PVR) of 3 Woods

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with pulmonary arterial hypertension and chronic thromboembolic pulmonary hypertension treated in Polish centres of pulmonary hypertension accredited by the National Health Fund
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Mortality | Since enrollment until at least 5 years.
  The number of patients who die during the follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Grzegorz Kopeć, MD, Phd, Principal Investigator — Krakowski Szpital Specjalistyczny im. Jana Pawła II
Locations (1):
- Krakowski Szpital Specjalistyczny im. Jana Pawła II, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Waligora M, Kurzyna M, Mularek-Kubzdela T, Skoczylas I, Chrzanowski L, Blaszczak P, Jaguszewski M, Kusmierczyk B, Ptaszynska K, Grzesk G, Mizia-Stec K, Malinowska E, Peregud-Pogorzelska M, Lewicka E, Tomaszewski M, Jachec W, Florczyk M, Mroczek E, Gasior Z, Pawlak A, Betkier-Lipinska K, Pruszczyk P, Widejko K, Zablocka W, Kopec G. Effects of beta-Blockers on the Outcomes in Patients With Pulmonary Arterial Hypertension Stratified by the Presence of Comorbid Conditions: A Multicenter Prospective Cohort Study: The Database of Pulmonary Hypertension in the Polish Population (BNP-PL). Chest. 2025 Apr;167(4):1171-1181. doi: 10.1016/j.chest.2024.10.051. Epub 2024 Nov 9. PMID 39528108
- [Derived] Kopec G, Dzikowska-Diduch O, Mroczek E, Mularek-Kubzdela T, Chrzanowski L, Skoczylas I, Tomaszewski M, Peregud-Pogorzelska M, Karasek D, Lewicka E, Jachec W, Gasior Z, Blaszczak P, Ptaszynska-Kopczynska K, Mizia-Stec K, Biederman A, Zielinski D, Przybylski R, Kedzierski P, Waligora M, Roik M, Grabka M, Orlowska J, Araszkiewicz A, Banaszkiewicz M, Slawek-Szmyt S, Darocha S, Magon W, Dabrowska-Kugacka A, Stepniewski J, Jonas K, Kaminski K, Kasprzak JD, Podolec P, Pruszczyk P, Torbicki A, Kurzyna M. Characteristics and outcomes of patients with chronic thromboembolic pulmonary hypertension in the era of modern therapeutic approaches: data from the Polish multicenter registry (BNP-PL). Ther Adv Chronic Dis. 2021 Mar 25;12:20406223211002961. doi: 10.1177/20406223211002961. eCollection 2021. PMID 33854746